CLINICAL TRIAL: NCT02670447
Title: Early Identification of Patients Presenting a First Psychotic Episode, Non Answering to First Line Support Strategies: A Multicentric Study
Brief Title: Early Identification of Patients Presenting a First Psychotic Episode, Non Answering to First Line Support Strategies
Acronym: PEPsy
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1508174; 2015-A01756-43 (Other: ANSM)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken for every patient to make toxicological tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First episode of psychosis patients: Patients with schizophrenia will be studied in this clinical trial, and that have never received anti-psychotic treatment. They will perform an MRI.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Magnetic Resonance Imagery will be performed on patients attempted by schizophrenia. The aim of this intervention is an early detection of the non-answering patients to the primary cares.
  Other Names: Magnetic Resonance Imagery

SUMMARY:
Researchers propose in this project to evaluate predictive factors of non response. It is defined by the lack of symptomatic remission at month 3, for patients presenting a first episode of psychosis. It will be performed on objective markers taken from imagery techniques. The link between evolution of these markers and clinical measures will be studied.

DETAILED DESCRIPTION:
Recently, radiological markers demonstrated a good capacity to discriminate first episode of psychosis patients, that will show a bad response to treatment. Furthermore, automatic learning methods were recently successfully applied to neurological data, but never for the first episode psychosis patients. These powerful methods are based on multivariate analyses allowing the prediction at an individual stage. The possibility to identify more precisely the population of non-answering patients would allow the adaptation of the support in first attention for these patients, and consequently to perform appropriate cares.

Researchers propose in this project to evaluate predictive factors of non response. It is defined by the lack of symptomatic remission at month 3, for patients presenting a first episode of psychosis. It will be performed on objective markers taken from imagery techniques. The link between evolution of these markers and clinical measures will be studied.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18-35 years
* member or beneficiary of a social security scheme,
* for women, appropriate contraception will be mandatory, as well as a negative pregnancy test,
* patients with a diagnosis of schizophrenia, schizoaffective disorder or schizophreniform disorder according to the DMS V
* having never received anti-psychotic treatment,
* followed in the hospital or outpatient,
* having given their written informed consent,
* that the physical examination revealed no significant clinical abnormalities

Exclusion Criteria:

* Female patients of childbearing period without effective contraception (oral, intramuscular hormonal, intrauterine device, or surgical);
* Patients pregnant or nursing;
* Presenting a serious somatic or neurological disease, especially Parkinson's disease, epilepsy, debilitating tardive dyskinesia, cardiovascular disease, severe liver or kidney;
* Featuring against-indication for an MRI; including: metallic foreign body eye or intracranial, pacemaker, heart valve, surgical clips, claustrophobia, large tattoo in the upper part of the body, not compatible with 3T MRI
* Having a history of alcohol or drug abuse in the past year;
* Participating in another clinical trial or being in an exclusion period of the previous protocol;
* Patients likely to exhibit aggressive behavior self according to the judgment of the investigators.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering of schizophrenia will be included in this study. They do not have ever taken anti-psychotic treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Score of the predictive value of the imagery markers. | Month 3
  Evaluate the predictive value for the imagery markers on the therapeutic non-answer at month 3 for patients presenting a first psychotic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Eric FAKRA, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - Chu Le Vinatier, Bron
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - HÔPITAL Edouard Herriot, Lyon
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No